CLINICAL TRIAL: NCT03434392
Title: QST Study: Predicting Treatment Response in Chronic Pancreatitis Using Quantitative Sensory Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Evans Phillips (Other)
Collaborators: Johns Hopkins University (Other); Aalborg University (Other)
Responsible Party: Sponsor-Investigator, Anna Evans Phillips, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO17060648
Record Dates: First submitted 2017-11-03; First posted 2018-02-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pancreatitis; Chronic Pain
Keywords: Chronic Pain; Chronic Pancreatitis; Sphincter of Oddi Dysfunction; Recurrent Acute Pancreatitis; Chronic Abdominal Pain; Functional Dyspepsia
MeSH Terms: conditions — Pancreatitis, Chronic; Chronic Pain; Sphincter of Oddi Dysfunction; Pancreatitis | interventions — Postsynaptic Potential Summation

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of four groups in parallel for the duration of the study based on prior clinical history.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Healthy Controls (Active Comparator): Subjects with no pancreatic disease and no abdominal pain.
  Subjects will undergo the following Interventions:
  Quantitative Sensory Test 1, Quantitative Sensory Test 2, and Quantitative Sensory Test 3, They will also fill out validated questionnaires.
  Interventions: Diagnostic Test: Quantitative Sensory Test 1; Diagnostic Test: Quantitative Sensory Test 2; Diagnostic Test: Quantitative Sensory Test 3
- Suspected CP (Active Comparator): Suspected Chronic Pancreatitis patients.
  Subjects will undergo the following Interventions:
  Quantitative Sensory Test 1, Quantitative Sensory Test 2, and Quantitative Sensory Test 3, They will also fill out validated questionnaires.
  Interventions: Diagnostic Test: Quantitative Sensory Test 1; Diagnostic Test: Quantitative Sensory Test 2; Diagnostic Test: Quantitative Sensory Test 3
- Definite CP (Active Comparator): Definite Chronic Pancreatitis patients.
  Subjects will undergo the following Interventions:
  Quantitative Sensory Test 1, Quantitative Sensory Test 2, and Quantitative Sensory Test 3, They will also fill out validated questionnaires.
  A subset of these patients who undergo endotherapy as per clinical recommendation from clinical provider independent of this study will be followed for 6 months after their clinical intervention for repeat Quantitative Sensory Test 1, Quantitative Sensory Test 2, and Quantitative Sensory Test 3 and questionnaires.
  Interventions: Diagnostic Test: Quantitative Sensory Test 1; Diagnostic Test: Quantitative Sensory Test 2; Diagnostic Test: Quantitative Sensory Test 3
- Sphincter of Oddi Dysfunction or Functional Dyspepsia (Active Comparator): Patients with Sphincter of Oddi Dysfunction Type 1 or Type 2, or who have a prior diagnosis of Functional Dyspepsia.
  Subjects will undergo the following Interventions:
  Quantitative Sensory Test 1, Quantitative Sensory Test 2, and Quantitative Sensory Test 3, They will also fill out validated questionnaires.
  Interventions: Diagnostic Test: Quantitative Sensory Test 1; Diagnostic Test: Quantitative Sensory Test 2; Diagnostic Test: Quantitative Sensory Test 3

INTERVENTIONS:
Diagnostic Test: Quantitative Sensory Test 1 — Subject will give pain rating (on Visual Analogue Scale (VAS) 0-10) of single as well as multiple stimulation with round-tip non-invasive pin-prick device. Difference is recorded as Temporal Summation Score.
  Other Names: Temporal Summation
Diagnostic Test: Quantitative Sensory Test 2 — Subject will state when they first detect pain and pain detection threshold in response to pressure administration with pressure algometer. Pressure threshold recorded in kilopascals(kP). Stimulation will be repeated in pancreatic and control dermatomes. Subject will then state pain tolerance threshold at same locations. Sensitization will be characterized by ratio of pancreatic vs. control dermatome scores.
  Other Names: Segmental v Systemic Sensitization
Diagnostic Test: Quantitative Sensory Test 3 — Subject will apply dominant hand to ice-chilled water bath (36F) for up to 2 minutes. Pain score (VAS 0-10) will be assessed each 10 seconds. Pain tolerance threshold (in kP) will be assessed with algometer on non-dominant thigh before and after water bath to determine change in threshold. Difference in pain tolerance recorded as Conditioned Pain Modulation Score.
  Other Names: Conditioned Pain Modulation

SUMMARY:
Quantitative Sensory Testing (QST) is a novel investigative technique used in other pain conditions to evaluate patterns of chronic pain, and in this study will be used to elucidate pain patterns in patients with Chronic Pancreatitis (CP). QST uses a specific series of standardized stimulations to map the pain system. QST has the potential to change and improve the treatment paradigm for patients with CP and may eventually be able to predict response to invasive CP therapies.

DETAILED DESCRIPTION:
In Chronic Pancreatitis (CP), clinical pain symptoms correlate poorly with pancreatic ductal morphology, response to endoscopic or surgical therapy is unpredictable, and the rationale for invasive therapies is often questioned. Quantitative sensory testing (QST) is a technique used to map the pain system based on the rationale that different neural pathways and networks can be explored using standardized stimulation and simultaneous recording of the evoked pain response by psychophysical and/or objective methods. In this study, the investigators aim to distinguish phenotypes characterized by segmental sensitization of the pancreatic viscerotome, and systemic sensitization with pathological central pain processing.

The investigators will perform QST on controls and CP subjects consisting of stimulation in several different dermatomes including pancreatic and control areas. All subjects will also answer standardized questionnaires assessing pain, depression, anxiety, and quality of life at baseline. Subjects undergoing endoscopic or surgical therapy will also undergo follow-up testing consisting of the same tests at 1, 3, and 6 months post-procedure for evaluation of changes in their pain profile.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with no pancreatic disease and no abdominal pain, or patients with a diagnosis of functional dyspepsia.

   * Subjects are 18 years or older in age
   * Subjects must be able to read and understand the study information.
   * Personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
   * Subject is willing and able to comply with the scheduled visits, questionnaires, treatment plan, and other study procedures.
2. Suspected CPs Inclusion Criteria

   * Subjects are 18 years or older in age
   * Subjects with a) Indeterminate CP (Cambridge 1 or 2 on CT scan or MRI/MRCP) who have abdominal pain without prior history of AP, or b) those with acute (AP) or recurrent acute pancreatitis (RAP) who have recovered from their attack(s) of AP, whose imaging studies are either normal or show changes consistent with Cambridge classification of 1 or 2, and they have ongoing abdominal pain. Both diabetic and non-diabetic subjects will be allowed to enter the study.
   * Subjects must be able to read and understand the study information.
   * Subjects must suffer from abdominal pain suspected to be pancreatic origin with an intensity above 3 on the visual analogue scale (VAS, where 0=no pain and 10= intolerable pain), and meet the criteria for chronic pain (pain ≥ 3 days per week for at least 3 months).
   * Personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
   * Subjects willing and able to comply with the scheduled visits, questionnaires, and other study procedures.
3. Definite Chronic Pancreatitis - Inclusion Criteria

   * Subjects are 18 years or older in age
   * Subjects will have a prior confirmed diagnosis of CP on CT scan or MRI/MRCP according to Cambridge Classification (grade 3 or 4). Both diabetic and non-diabetic subjects will be allowed to enter the study.
   * Subjects must be able to read and understand the study information.
   * Personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
   * Subjects willing and able to comply with the scheduled visits, questionnaires, and other study procedures.
4. Sphincter of Oddi Dysfunction (SOD) Type 1 or Type 2 Inclusion Criteria

   * Subjects are 18 years or older in age
   * Subjects have prior diagnosis of Type 1 or Type 2 Sphincter of Oddi Dysfunction (subjects with biliary pain accompanied by biochemical features of transient biliary tract obstruction including elevated transaminases, alkaline phosphatase, or conjugated bilirubin; may also be accompanied by biliary or pancreatic ductal dilation on imaging)
   * Subjects must be able to read and understand the study information.
   * Personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
   * Subjects willing and able to comply with the scheduled visits, questionnaires, and other study procedures.

Exclusion Criteria:

1. Subjects with no pancreatic disease and no abdominal pain, or patients with a diagnosis of functional dyspepsia.

   * Subjects with evidence or history of medical or surgical disease of importance for this study as judged by investigator.
   * Subjects suffering from painful conditions that make them unable to distinguish the pain associated with CP from chronic pain of other origins.
   * Subjects with known pregnancy at the time of enrolment.
   * Subjects who have previously undergone surgical intervention on their pancreas.
2. Suspected CPs Exclusion Criteria

   * Subjects with evidence or history of medical or surgical disease of importance for this study as judged by investigator.
   * Subjects suffering from painful conditions other than pancreatitis or SOD type 1 or 2 that make them unable to distinguish the pain associated with pancreatitis or SOD from chronic pain of other origins.
   * Subjects with known pregnancy at the time of enrolment.
   * Subjects who have previously undergone surgical intervention on their pancreas.
3. Definite Chronic Pancreatitis Exclusion Criteria

   * Subjects with evidence or history of medical or surgical disease of importance for this study as judged by investigator.
   * Subjects suffering from painful conditions other than pancreatitis or SOD type 1 or 2 that make them unable to distinguish the pain associated with pancreatitis or SOD from chronic pain of other origins.
   * Subjects with known pregnancy at the time of enrolment.
   * Subjects who have previously undergone surgical intervention on their pancreas.
4. Sphincter of Oddi Dysfunction (SOD) Type 1 or Type 2 Exclusion Criteria

   * Subjects with evidence or history of medical or surgical disease of importance for this study as judged by investigator.
   * Subjects suffering from painful conditions other than pancreatitis or SOD that make them unable to distinguish the pain associated with pancreatitis or SOD from chronic pain of other origins.
   * Subjects with known pregnancy at the time of enrolment.
   * Subjects who have previously undergone surgical intervention on their pancreas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-10-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Pattern Assessment as assessed by the combination of Temporal Summation score, Sensitization score, and Conditioned Pain Modulation score | One-time baseline testing
  Assignment to one of four groups (Segmental Sensitization, Systemic Sensitization, Impaired Conditioned Pain Modulation, or Other) based on combination of patient-reported pain symptoms. Temporal summation pain symptoms are measured on visual analogue scales which are measured from 0 (minimum) to 10 (maximum). 10 on this scale indicates worse pain; 0 indicates no pain. Sensitization scores are measured via patient reported thresholds in kilopascals. Conditioned Pain modulation is measured also via patient reported threshold in kilopascals.

SECONDARY OUTCOMES:
Change in Mean Pain score | 90 days
  In Definite CP Patients undergoing endotherapy as part of regular clinical care, assessment of mean pain level for 7 days prior to endotherapy will be assessed immediately pre-procedure and again at 90 days post-procedure. A pain reduction of >30% in 90 days after procedure will be characterized as positive response to procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Evans-Phillips, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Johns Hopkins Medical Institutions, Baltimore, Maryland
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phillips AE, Faghih M, Singh VK, Bick B, Yadav D, Drewes AM, Olesen SS. Widespread Hyperalgesia by Pancreatic Quantitative Sensory Testing Is Associated With Reduced Pain Response in Chronic Pancreatitis. Pancreas. 2023 Apr 1;52(4):e257-e258. doi: 10.1097/MPA.0000000000002247. Epub 2023 Nov 13. No abstract available. PMID 37967828
- [Derived] Phillips AE, Faghih M, Singh VK, Olesen SS, Kuhlmann L, Novovic S, Bick B, Hart PA, Ramsey ML, Talukdar R, Garg PK, Yadav D, Drewes AM; Pancreatic Quantitative Sensory Testing (P-QST) Consortium. Rationale for and Development of the Pancreatic Quantitative Sensory Testing Consortium to Study Pain in Chronic Pancreatitis. Pancreas. 2021 Oct 1;50(9):1298-1304. doi: 10.1097/MPA.0000000000001912. PMID 34860815
- [Derived] Olesen SS, Phillips AE, Faghih M, Kuhlmann L, Steinkohl E, Frokjaer JB, Bick BL, Ramsey ML, Hart PA, Garg PK, Singh VK, Yadav D, Drewes AM; Pancreatic Quantitative Sensory Testing (P-QST) Consortium. Overlap and cumulative effects of pancreatic duct obstruction, abnormal pain processing and psychological distress on patient-reported outcomes in chronic pancreatitis. Gut. 2022 Dec;71(12):2518-2525. doi: 10.1136/gutjnl-2021-325855. Epub 2021 Oct 21. PMID 34675068
- [Derived] Phillips AE, Faghih M, Kuhlmann L, Larsen IM, Drewes AM, Singh VK, Yadav D, Olesen SS; Pancreatic Quantitative Sensory Testing (P-QST) Consortium. A clinically feasible method for the assessment and characterization of pain in patients with chronic pancreatitis. Pancreatology. 2020 Jan;20(1):25-34. doi: 10.1016/j.pan.2019.11.007. Epub 2019 Nov 20. PMID 31787527

DOCUMENTS (1):
  • Study Protocol (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT03434392/Prot_000.pdf